CLINICAL TRIAL: NCT06483256
Title: Evaluation of Clinical and Radiographic Findings in Patients Treated Surgically for Biceps Long Head Injury
Acronym: Artro-Bic
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Enrico Guerra, Principal investigator, Istituto Ortopedico Rizzoli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Artro-Bic
Record Dates: First submitted 2024-06-21; First posted 2024-07-03 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Bicep Tendon Rupture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- radiographic control (Other): Standard AP and LL X-Rays of the affected elbow
  Interventions: Diagnostic Test: radiographic control

INTERVENTIONS:
Diagnostic Test: radiographic control — Radiographic study with standard projections (AP and LL) is used to assess any signs of anchor loosening and/or presence of heterotopic ossifications (which can restrict movement and is one of the main complications).

SUMMARY:
This is an interventional, single-center study with clinical and radiographic evaluation, at follow-up of at least 2 years, of patients treated surgically with arthroscopy-assisted distal biceps tendon repair at the Rizzoli Orthopaedic Institute. The study consists of 2 phases (Identification of includable patients, Follow-up visit:

* identification by trained medical staff of subjects who meet the study inclusion criteria
* Patients, after signing informed consent, will be evaluated clinically and radiographically by radiography in lateral and anteroposterior projection at the follow-up visit by specialized medical personnel. A clinical examination will be performed, with subjective and objective evaluation questionnaires administered, and a strength assessment of the operated limb and contralateral limb will be performed using specific dynamometers on the same date as the radiography is performed at the Rizzoli Orthopedic Institute. The radiographic study with standard projections (AP and LL) is used to evaluate any signs of anchor loosening and/or presence of heterotopic ossifications (which can limit movement and represent one of the main complications).

Study-specific radiographs will be performed on the same day as the outpatient clinical evaluation in consultation with the Radiology Service Manager.

DETAILED DESCRIPTION:
This is an interventional, single-center study with clinical and radiographic evaluation, at follow-up of at least 2 years, of patients treated surgically with arthroscopy-assisted distal biceps tendon repair at the Rizzoli Orthopaedic Institute. The study consists of 2 phases (Identification of includable patients, Follow-up visit:

identification by trained medical staff of subjects who meet the study inclusion criteria Patients, after signing informed consent, will be evaluated clinically and radiographically by radiography in lateral and anteroposterior projection at the follow-up visit by specialized medical personnel. A clinical examination will be performed, with subjective and objective evaluation questionnaires administered, and a strength assessment of the operated limb and contralateral limb will be performed using specific dynamometers on the same date as the radiography is performed at the Rizzoli Orthopedic Institute. The radiographic study with standard projections (AP and LL) is used to evaluate any signs of anchor loosening and/or presence of heterotopic ossifications (which can limit movement and represent one of the main complications).

Study-specific radiographs will be performed on the same day as the outpatient clinical evaluation in consultation with the Radiology Service Manager.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 at the time of distal biceps tendon repair surgery
* Surgery performed within 30 days of injury
* Patients treated surgically for distal biceps tendon injury by arthroscopy-assisted technique at the Shoulder-Elbow Department of the Rizzoli Orthopedic Institute from January 01, 2017 to December 31, 2022.

Exclusion Criteria:

* < 18 years old at the time of surgery
* Patients who have presented non-surgery-related problems to the operated limb in the years following surgery such as fractures or subsequent episodes of tendon injury.
* Patients treated for distal biceps tendon injury by different surgical techniques

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Mayo elbow performance score | baseline (post surgery)
  It is currently considered the gold standard for objective measurement of elbow performance because of the immediacy of the results and its practicality of use. It assesses the presence of pain with a score from 0 to 45, Range of Motion with a score from 0 to 20, elbow stability with a score from 0 to 10, and the ability to perform 5 daily activities (combing, eating, personal hygiene, dressing, and putting on shoes) to each of which 5 points are assigned. It gives a result from 0 to 100 where results above 90 are defined as excellent, results between 75 and 89 are defined as good, between 60 and 74 are defined as sufficient and below 59 as poor.

SECONDARY OUTCOMES:
Disabilities of arm, shoulder and hand score | baseline (post surgery)
  is the most widely used score in the literature for objective assessment of upper limb function. Unlike MEPS, it is not a specific score for elbow pathology, but is widely used in the study of musculoskeletal disorders of other joints such as shoulder, wrist or in hand performance. The score is calculated by administering 30 items to the patient thus obtaining a score ranging from 0 (no disability) to 100 (maximum disability).
force evaluations with dynamometers | baseline (post surgery)
  Force assessments will be made with dynamometers for forearm supination and elbow flexion by going to compare the strength of the operated limb with that of the contralateral limb in order to obtain a ratio that allows comparison between patients
complications and reinterventions | baseline (post surgery)
  Questions will also be asked about possible complications and re-interventions, re-ruptures as well as return to pre-injury, pre-surgery daily activities, level of function achieved after the surgical procedure and maintenance of the same over time.
patient satisfaction | baseline (post surgery)
  A survey will be used to assest the patient satisfaction with their post-surgery recovery status. The patient will choose from 5 options to assest his general response to the surgery to see if it's better, worst or if nothing changed.
radiography | baseline (post surgery)
  Radiography (X-ray) to document signs of indirect anchor mobilization and formation of heterotopic ossifications.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Srinivasan RC, Pederson WC, Morrey BF. Distal Biceps Tendon Repair and Reconstruction. J Hand Surg Am. 2020 Jan;45(1):48-56. doi: 10.1016/j.jhsa.2019.09.014. PMID 31901332
- [Background] Schmidt CC, Madonna TJ, Vaudreuil N, Brown BT, Liu SY, Delserro S, Smolinski MP, Styron J, Smolinski PJ, Miller MC. The effect of tendon rotation on distal biceps repair. JSES Open Access. 2019 Sep 11;3(3):225-231. doi: 10.1016/j.jses.2019.06.001. eCollection 2019 Oct. PMID 31709367